CLINICAL TRIAL: NCT00520754
Title: The Efficacy and Safety of Levocetirizine Dihydrochloride Oral Drops Given 0.125 mg/kg b.i.d. During 90 Days in the Treatment of Recurrent Cough Associated With Other Allergic Symptoms, e.g. Wheezing, in Children Aged 1-2 Years.
Brief Title: Efficacy and Safety of Levocetirizine for Treatment of Recurrent Cough Associated With Other Allergic Symptoms in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A00315
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2009-09

CONDITIONS: Cough
Keywords: levocetirizine dihydrochloride Xyzal tablets
MeSH Terms: conditions — Cough | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levocetirizine dihydrochloride

SUMMARY:
Efficacy and Safety of Levocetirizine for Treatment of Recurrent Cough Associated With Other Allergic Symptoms in Children

ELIGIBILITY:
Inclusion Criteria:

* infants from 2 to 24 months both inclusive
* suffering from recurrent cough associated with other allergic symptoms
* hospitalized for respiratory or allergy related problems
* laboratory results within normal ranges
* height and weight between percentile 5 and 95

Exclusion Criteria:

* having taken any of the disallowed medication
* suffering form any disorder
* history of sleep apnea
* having concomitant chronic disease
* known relevant renal, hepatic, cardiac or metabolism dysfunction
* known alcohol or drug addiction, severe psychiatric disease for the parent/guardian

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2001-12; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
The efficacy based on daily record cards recordings | 90 days

SECONDARY OUTCOMES:
Safety and pharmacokinetics at 90 days; skin reactivity

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Cranswick N, Turzikova J, Fuchs M, Hulhoven R. Levocetirizine in 1-2 year old children: pharmacokinetic and pharmacodynamic profile. Int J Clin Pharmacol Ther. 2005 Apr;43(4):172-7. doi: 10.5414/cpp43172. PMID 15966463